CLINICAL TRIAL: NCT02861079
Title: Compare Prostaglandin E2 Against to Combined Use of Transcervical Foley Catheter Balloon With Vaginal Prostaglandin E2 for Induction of Labor at Term: A Randomized Study
Brief Title: Combined Foley Catheter Balloon and PGE2 Vaginal Ovule for Induction of Labor at Term: A Randomized Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, medical doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Unfavorable Cervix, Cervical Ripening
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propess with Foley balloon catheter (Experimental): 10 mg PGE2 vaginal ovul will be inserted to the posterior fornix and an 18-F Foley catheter which filling with 30 mL of saline solution will be placed into the cervix
  Interventions: Device: Foley catheter; Drug: PGE2
- Propess vaginal ovule (Active Comparator): 10 mg PGE2 vaginal ovule will be inserted to the posterior fornix
  Interventions: Drug: PGE2

INTERVENTIONS:
Device: Foley catheter — An 18-F Foley catheter will insert into the endocervical canal and the balloon will fill with 30 mL of saline solution.
  Arms: Propess with Foley balloon catheter
Drug: PGE2 — 10 mg PGE2 vaginal ovul (Propess,Ferring®) will place high into the posterior vaginal fornix.
  Other Names: propess

SUMMARY:
This study evaluates the addition of transcervical Foley catheter balloon and vaginal prostaglandin E2 in induction of labor at term. Half of participants will be used combine transcervical Foley catheter balloon and vaginal prostaglandin E2, while the other half will be used alone vaginal prostaglandin E2.

DETAILED DESCRIPTION:
An unfavorable cervix during induction decreases the success rate of labor induction and vaginal delivery. Therefore it is required to apply cervical ripening methods for unfavorable cervices. Application of transcervical Foley catheter is an effective mechanical method and has the advantages of lower cost and lowest rate of fetal heart rate changes due to tachysystole compared with PGE1 and PGE2. Despite the advantages of mechanical methods, PGE1 and PGE2 are reported to be more effective than mechanical methods to achieve vaginal delivery within 24 hours. Although there are a lot of studies comparing PGE1, PGE2 and transcervical Foley balloon catheter separately and PGE1 combined with transcervical Foley balloon catheter, less is known about combined usage of PGE2 and transcervical Foley balloon catheter.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy,
2. gestational age ≥37 weeks,
3. intact membranes,
4. cephalic presentation,
5. bishop score ≤5,
6. had obstetrical indications for induction of labor,
7. had less than three uterine contractions in every 10 minutes. -

Exclusion Criteria:

1. Patients who had contraindications for vaginal delivery,
2. previous uterine surgery,
3. fetal malpresentation,
4. multifetal pregnancy,
5. more than three contractions in 10 minutes,
6. contraindications to prostaglandins,
7. a category II or III fetal heart rate pattern,
8. anomalous fetus,
9. fetal demise
10. women with immediate delivery indications -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
induction-to- delivery time | the length of time between the beginning of induction and the end of labor
  the length of time between the beginning of induction and the end of labor

SECONDARY OUTCOMES:
induction-to-active phase of labor time | the length of time between the beginning of induction and the onset of labor
  the length of time between the beginning of induction and the onset of labor

CONTACTS AND LOCATIONS:
Overall Officials: ahmet eser, M.D., Study Director — Zeynep Kamil Maternity and Children's Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey
Locations (1):
- Zeynep Kamil Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Du C, Liu Y, Liu Y, Ding H, Zhang R, Tan J. Double-balloon catheter vs. dinoprostone vaginal insert for induction of labor with an unfavorable cervix. Arch Gynecol Obstet. 2015 Jun;291(6):1221-7. doi: 10.1007/s00404-014-3547-3. Epub 2014 Nov 19. PMID 25408273
- [Result] Dalui R, Suri V, Ray P, Gupta I. Comparison of extraamniotic Foley catheter and intracervical prostaglandin E gel for preinduction cervical ripening. Acta Obstet Gynecol Scand. 2005 Apr;84(4):362-7. doi: 10.1111/j.0001-6349.2005.00662.x. PMID 15762966
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264